CLINICAL TRIAL: NCT02899026
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Sirukumab in Subjects With Polymyalgia Rheumatica
Brief Title: Efficacy and Safety Study of Sirukumab in Subjects With Polymyalgia Rheumatica
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: GSK decision to return rights to sirukumab to Janssen and discontinue sirukumab development in polymyalgia rheumatica.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205012
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Polymyalgia Rheumatica
Keywords: Glucocorticosteroids; Sirukumab; Prednisone; Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — sirukumab; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Sirukumab 100 mg SC + prednisone (6-week taper) (Experimental): Eligible subjects will receive blinded Sirukumab 100 mg subcutaneously (SC) every 2 weeks (q2w) for 52 weeks plus a 6-week oral prednisone taper regimen
  Interventions: Drug: Sirukumab; Drug: Prednisone /Prednisone placebo
- Part A: Sirukumab 50 mg SC + prednisone (6-week taper) (Experimental): Eligible subjects will receive blinded Sirukumab 50 mg SC q4w (with placebo SC injections q2w between sirukumab injections) for 52 weeks plus a 6-week oral prednisone taper regimen
  Interventions: Drug: Sirukumab; Drug: Placebo to match sirukumab; Drug: Prednisone /Prednisone placebo
- Part A: Placebo SC + prednisone (52 week taper) (Placebo Comparator): Eligible subjects will receive blinded placebo SC q2w for 52 weeks plus a blinded 52-week oral prednisone taper
  Interventions: Drug: Placebo to match sirukumab; Drug: Prednisone /Prednisone placebo

INTERVENTIONS:
Drug: Sirukumab — Sirukumab will be provided as 1 millilitre (mL) Pre-filled Syringe (PFS), containing 100 mg/mL or 50 mg/mL of sirukumab, fitted with a spring-powered, disposable autoinjector device for single use SC administration of liquid biologic drug
  Arms: Part A: Sirukumab 100 mg SC + prednisone (6-week taper); Part A: Sirukumab 50 mg SC + prednisone (6-week taper)
Drug: Placebo to match sirukumab — Placebo to match sirukumab will be provided as 1.0 mL PFS fitted with a spring-powered, disposable autoinjector device for single use SC administration of liquid biologic drug
  Arms: Part A: Placebo SC + prednisone (52 week taper); Part A: Sirukumab 50 mg SC + prednisone (6-week taper)
Drug: Prednisone /Prednisone placebo — Prednisone will be provided as tablets with dosage level up to 20 mg/day. All subjects will receive 20 mg prednisone at Baseline (Randomization) and follow predefined taper regimen (6 weeks or 52 weeks) based on treatment assignment. Placebo to match prednisone will be provided as tablets

SUMMARY:
Sirukumab is a human anti-IL-6 monoclonal antibody that selectively binds to the cytokine with high affinity that may have therapeutic benefit in the treatment of polymyalgia rheumatica (PMR) by interrupting multiple pathogenic pathways. Sirukumab inhibits IL-6-mediated signal transducer and activator of transcription 3 (STAT3) phosphorylation, resulting in the inhibition of the biological effect of IL-6. This study will evaluate the efficacy and safety of sirukumab to characterize the benefit-to-risk profile of sirukumab in the treatment of active PMR. The study will be conducted in 2 parts (Part A and Part B) and consists of the following phases: Screening phase, Part A: 52-week double-blind treatment phase, Part B: 52-week extension phase with no study drug administration and a 16-week follow-up phase if applicable.

Approximately 150 subjects with a diagnosis of PMR and active disease within 6 weeks of baseline will be randomized into Part A, the 52-week double-blind treatment phase, to receive one of two doses of sirukumab or placebo, each in addition to a pre-specified prednisone taper. The efficacy and safety of sirukumab in sustaining remission will be assessed at Week 52. Subjects completing Part A of the study who are in clinical remission will be eligible to enter Part B, the 52-week extension phase, designed to investigate the long-term maintenance of remission and safety following cessation of sirukumab treatment and to assess long-term corticosteroid use. Subjects will need to have follow-up safety evaluations for at least 16 weeks after receiving the last dose of study drug, applicable for those who have withdrawn prematurely from the study or who have completed Part A but are not eligible for Part B.

ELIGIBILITY:
Inclusion Criteria:

* Age >=50 years
* Diagnosis of PMR based on the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) 2012 provisional PMR classification criteria, that is, at the time of PMR diagnosis, subjects should be aged 50 years or older, presenting with new-onset (<12 weeks of diagnosis) bilateral shoulder pain and abnormal acute-phase response, and are required to score 4 or more on the following criteria for the diagnosis of PMR: Morning stiffness duration >45 minutes (2 points) or Hip pain or limited range of motion (1 point) or Absence of rheumatic factor (RF) or anti-citrullinated protein antibody (ACPA) (2 points) or Absence of other joint involvement (1 point).
* Active PMR within 6 weeks of randomization where active disease is defined by an ESR >=30 millimeter (mm)/hour (hr) or CRP >=1 mg/dL within 6 weeks of randomization AND the presence of at least one of the following at screening (within 6 weeks of randomization): Unequivocal symptoms of PMR, defined as shoulder and/or hip girdle pain associated with inflammatory stiffness or Other features judged by the clinician investigator to be consistent with PMR or PMR flares (e.g. fever of unknown origin).
* Receiving oral prednisone 0-25 mg once daily (or equivalent) for PMR treatment at screening. Dosage of oral prednisone or equivalent, during the screening period can remain constant or be adjusted within the range of 0-25 mg prednisone equivalent based on investigator's discretion.
* Willing and able to receive treatment with oral prednisone 20 mg once daily at randomization and undergo a pre-defined blinded prednisone taper.
* No evidence of active or latent infection with Mycobacterium tuberculosis (TB)
* Be able to read, understand, and complete study questionnaires.
* Male and female subjects, where male subjects with female partners of child bearing potential must comply with the contraception requirements and not to donate sperm from the time of first dose of study medication until 4 months after the last dose of study medication. A female subject of child bearing potential must comply with contraception requirements.

Exclusion Criteria:

* Features consistent with atypical PMR according to the investigator's clinical judgment. Investigators are encouraged to discuss with the medical monitor when there are questions regarding excluding subjects with atypical PMR. Atypical features or features that increase the likelihood of a non-PMR diagnosis may include some or all of the following: Age <60 years; Chronic onset (>2 months) at time of diagnosis; Lack of shoulder involvement; lack of inflammatory stiffness; prominent systemic features, weight loss, night pain, neurological signs; features of other rheumatic disease; Normal or extremely high acute-phase response; AND treatment dilemmas such as incomplete, poorly sustained or non-response to GCs, inability to reduce GCs, contraindications to GC therapy, the need for prolonged GC therapy (>2 years).
* History or current diagnosis of Giant Cell Arteritis (GCA), or Large Vessel Vasculitis (LVV). If GCA/LVV is suspected, this should be ruled out by ultrasound or other imaging techniques (example. fluorodeoxy-glucose positron emission tomography) prior to entering the study.
* Maintained on GCs for 2 years or more prior to Screening.
* Other inflammatory rheumatic diseases with the exception of gout controlled on stable suppressive therapy and without flares for at least 2 years prior to screening and expected to remain on this therapy for the duration of the study.
* Recent (within the past 12 weeks) or planned major surgery that would impact on study procedures or assessments.
* Organ transplantation recipients (except corneas within 3 months prior to randomization visit).
* Requires continued or repeated use of systemic GCs for conditions other than PMR.
* Evidence of serious concomitant disease, which in the opinion of the investigator makes the subject unsuitable for participation in the study for either safety or efficacy.
* Major ischemic event within 12 weeks of screening.
* At screening, marked prolongation of corrected QT interval (QTc) > 450 millisecond (msec) [QTc by Bazett's formula (QTcB) or QTc by Fridericia's formula (QTcF)] or QTc > 480 msec in subjects with Bundle Branch Block. History of Torsade de Pointes, family history of long QT syndrome, history of second or third degree heart block.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of or current active diverticulitis, inflammatory bowel disease, or other symptomatic gastro intestinal (GI) tract condition that might predispose to bowel perforation.
* History of known demyelinating diseases such as multiple sclerosis or optic neuritis.
* Active infections, or history of recurrent infections or required management of acute or chronic infections, as follows: currently on any suppressive therapy for a chronic infection and History or suspicion of chronic infection (e.g. joint infection) OR Hospitalization for treatment of infection within 60 days of the randomization visit OR Use of parenteral (intravenous [IV] or intramuscular [IM]) antimicrobials (antibacterials, antivirals, antifungals, or antiparasitic agents) within 60 days of randomization or oral antimicrobials within 30 days of randomization.
* Primary or secondary immunodeficiency.
* Human immunodeficiency syndrome (HIV) infection, hepatitis C.
* Hepatitis B infection
* Active malignancy or history of malignancy within previous 5 years.
* Any other autoimmune disease.
* Uncontrolled thyroid disease.
* Uncontrolled psychiatric or emotional disorder.
* Current history of suicidal ideation or past history of suicide attempt.
* Has received prior treatment with any of the following: Systemic immunosuppressives within 4 weeks of randomization; Systemic GCs for conditions other than PMR within 8 weeks of randomization; Biologic agents targeted at reducing Tumor necrosis factor (TNF) alpha within 4-8 weeks of randomization, depending on the agent; B-cell depleting agents (e.g., rituximab) within 12 months prior to baseline or longer if B cell counts have not returned to the normal range or baseline levels; Any prior use of tocilizumab or other anti-IL-6 agents, Cytotoxic drugs such as cyclophosphamide, chlorambucil, nitrogen mustard, or other alkylating agents, Abatacept and Tofacitinib; Methotrexate use within 2 weeks of randomization; Methylprednisolone > 100 mg/day IV (or equivalent) within 8 weeks of randomization.
* Has received, or is expected to receive, any live virus or bacterial vaccination within 3 months of randomization, during the study, or within 4 months after the last administration of study treatment. Have had a Bacille Calmette Guérin (BCG) vaccination within 12 months of screening.
* Has received an investigational drug (including investigational vaccines) or used an investigational medical device within 3 months or 5 half-lives, whichever is longer, before randomization.
* History of drug abuse, alcohol abuse within 3 years prior to screening.
* History of severe allergic reactions to monoclonal antibodies, human proteins, or excipients.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* Laboratory abnormalities at screening
* A female subject who is pregnant or lactating.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2020-08-26 (Estimated); Study Completion 2021-08-26 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects in sustained | Week (wk) 52
  Sustained remission at Week 52 is defined as having achieved all of the following: Remission by Week 12; Absence of disease flare following remission at Week 12 through Week 52; Completion of the assigned prednisone taper protocol; No requirement for rescue therapy at any time through Week 52. One flare before Week 12 is permitted if it can be successfully treated with a 5 mg/day prednisone add-on taper regimen in addition to the predefined taper schedule providing all other sustained remission criteria are met.

SECONDARY OUTCOMES:
Part A: Cumulative prednisone dose at Week 52 | Week 52
  Cumulative prednisone dose at Week 52 (Part A)
Part A&B: Cumulative prednisone dose over time | Over 104 weeks
  Cumulative prednisone dose over time
Part A&B: Proportion of subjects in sustained remission | Week 12 to Week 52 (Part A) and to Week 104 (Part B)
  Subjects with sustained disease remission will be evaluated
Part A&B: Proportion of subjects in remission while on a daily prednisone dose of 5mg | Week 52 (Part A) and Week 76 (Part B)
  Subjects in remission while on a daily prednisone dose of 5mg will be evaluated
Part B: Proportion of subjects in remission while off prednisone | Week 76 (Part B)
  Proportion of subjects in remission while off prednisone at baseline of Part B and who remain off prednisone during the first 24 weeks of Part B
Part A&B: Time to first PMR disease flare | 52 weeks (Part A) and 104 weeks (Part B)
  Time to first PMR flare after remission
Part A&B: Number of PMR disease flares per subject over time | 52 weeks (Part A) and 104 weeks (Part B)
  PMR disease flare over time
Part A: Change in PMR-activity score (AS) | Week 12 and 52
  Change in PMR-AS score from baseline to Week 12 and 52
Part A: Proportion of subjects meeting PMR-AS remission criteria of <1.5 | Week 12 and 52
  Subjects withng PMR-AS remission criteria of <1.5
Part A&B: Incidence of adverse events (AEs) and Serious AEs (SAEs) | 52 weeks (Part A) and 104 weeks (Part B)
  All AEs and SAEs will be reported
Part A: Incidence of GC-related AEs | 52 weeks
  GC-related AEs will be reported
Part A&B: Vital sign assessment as measure of safety | Baseline (Week 0) to Week 52 (Part A) and Week 104 (Part B)
  Vital sign assessment includes systolic and diastolic blood pressure, pulse rate and body temperature
Part A&B: Number of subjects having abnormal hematology parameters as a measure of safety | Baseline (Week 0) to Week 52 (Part A) and Week 104 (Part B)
  Blood samples will be collected to measure hematological parameters such as platelet count, red blood cell (RBC) count, hemoglobin, hematocrit, white blood cell (WBC) count (including neutrophil count, lymphocyte count, monocyte count, eosinophil count and basophils count).
Part A&B: Number of subjects having abnormal clinical chemistry parameters as a measure of safety | Baseline (Week 0) to Week 52 (Part A) and Week 104 (Part B)
  Blood samples will be collected to measure serum chemistry parameters such as sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, glucose aspartate transaminase, alanine transaminase, alkaline phosphatase, calcium, phosphate, albumin, total protein, direct, indirect and total bilirubin
Part A&B: Assessment of quality of life using the 36-item Short Form Health Survey version 2 (SF-36v2) (acute) | 52 weeks (Part A) and 104 weeks (Part B)
  Patient report of quality of life
Part A&B: Functional Assessment of Chronic Illness Therapy (FACIT )-Fatigue | 52 weeks (Part A) and 104 weeks (Part B)
  Patient report of elements of fatigue
Part A&B: Assessment of pain | 52 weeks (Part A) and 104 weeks (Part B)
  Pain assessed by patient reported rating on a numeric rating scale from 0 to 10
Part A&B: Assessment of steroid impact | 52 weeks (Part A) and 104 weeks (Part B)
  Patient assessment of the side effects and impact of steroids on PMR symptoms over time
Part A&B: Modified Health Assessment Questionnaire (MHAQ) | 52 weeks (Part A) and 104 weeks (Part B)
  Patient reported outcome of disease-related disability, discomfort, and quality of life
Part A&B: Assessment of Patient Global Impression of Change (PGIC) | 52 weeks (Part A) and 104 weeks (Part B)
  Estimate of the magnitude of patient response to treatment at different time points by patient report
Part A&B: Patient Global Assessment of Disease Activity (PtGA) | 52 weeks (Part A) and 104 weeks (Part B)
  Patient report of PMR disease activity
Part A&B: Duration of Morning Stiffness | 52 weeks (Part A) and 104 weeks (Part B)
  Patient report of the duration of morning stiffness
Part A&B: Physician Global Assessment of Disease Activity (PhGA) | 52 weeks (Part A) and 104 weeks (Part B)
  Physician assessment of PMR disease activity on a scale of 0-100
Part A&B: Pharmacokinetics: Serum concentrations of sirukumab | 68 weeks
  Blood samples for Pharmacokinetic (PK) analysis of sirukumab serum concentrations will be collected at Baseline, wk 4, wk 8, wk 12, wk 16, wk 24, wk 36 and wk 52 in Part A; and at wk 60 and wk 68 (Part B)
Part A&B: Serum anti-sirukumab antibodies | 68 weeks
  Blood samples for antibodies analysis of sirukumab will be collected at Baseline, wk 24 and wk 52 in Part A; and at wk 68 in Part B

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: No